CLINICAL TRIAL: NCT04611555
Title: Implementation of the International Classification of Functioning, Disability and Health Model in Cochlear Implant Recipients: a Multi-center Prospective Follow-up Cohort Study
Brief Title: ICF in Cochlear Implant Users
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Collaborators: World Hearing Centre (Unknown); Hospital Universitario La Paz (Other); Fiona Stanley Hospital (Other); Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, Griet Mertens, Prof., University Hospital, Antwerp
Other Study IDs: B3002020000137
Record Dates: First submitted 2020-10-20; First posted 2020-11-02 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Hearing Loss
Keywords: Cochlear Implantation; International Classification of Functioning, Disability and Health
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CI users

SUMMARY:
The current project proposes a multi-center prospective follow-up cohort study aiming to realize an international framework to classify human functioning and disability in Cochlear Implant (CI) recipients using a standardized ICF framework. For this, ICF qualifiers which denote the magnitude of the level of health or severity of the problem will be quantified to enable comparison of data across countries and health-care disciplines. Adult subjects (≥18 years old) eligible for cochlear implantation, considering the local criteria of reimbursement, will be assessed one month preoperatively and six months post the activation of the speech processor using three audiological examinations, evaluating the participants' localization abilities, speech recognition and hearing thresholds, and six questionnaires, each evaluating different aspects of daily life functioning and disability in hearing-impaired persons.

ELIGIBILITY:
Inclusion Criteria:

1. General

   * Adults aged 18 years or older with postlingual HL
   * Signed and dated informed consent, informed permission and/or minors assent.
   * Willingness to participate in evaluations, test sessions, and medical follow-up sessions as defined in the protocol.
   * Physical and mental competence to participate in fitting of the device and follow-up sessions as defined in the protocol.
   * Fluency in the language of the implanting centre.
2. Audiological

   * Completion of hearing assessment battery showing suitability of the CI candidates.
   * Compliance with cochlear implant candidate selection criteria of the implanting centre.
   * First cochlear implantation
3. Medical

   * Patent cochlea, as evidenced by High-resolution computed tomography (HRCT) and/or Magnetic Resonance Imaging (MRI).

Exclusion Criteria:

1. General

   * Re-implantation of the cochlear implant
   * No motivation to participate in the study and/or unreasonable expectations.
2. Medical

   * Presence of contra-indications for surgery in general and cochlear implantation in particular.
   * Presence of central auditory lesions.
   * Autoimmune disease, meningitis or ossification of the cochlea.
   * Radiological evaluation indicating malformation or obstruction of the cochlea.
   * Unstable psychological status.
   * Any disorder that may relate to an increased risk of skin flap problems
   * Having received chemotherapy
   * Be a burn victim
3. Use of one of the following electrodes for implantation

   * Compressed
   * Split
   * Any type of custom made electrodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult subjects (≥18 years old) eligible for cochlear implantation, considering the local criteria of reimbursement.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change in Work Rehabilitation Questionnaire (WORQ) | One month preoperatively and six months post the activation of the speech processor
  The WORQ was divided into two sections. Section one contains 18 sociodemographic and work-related questions regarding the four environmental categories from the brief ICF Core Set. The six categories from activities and participation that describe vocational education or work situations namely were also included in section one. In the main section of WORQ, 36 questions were phrased representing 34 categories. The WORQ has been revised to match the core needs of the cochlear implant ICF codes. The revised version includes 4 items in the first section and 14 items in the main section, taking less than 5 minutes to complete.
Change in Abbreviated Profile of Hearing Aid Benefit (APHAB) | One month preoperatively and six months post the activation of the speech processor
  The APHAB is a 24-item questionnaire derived from the original 66-item Profile of Hearing Aid Benefit. The self-assessment instrument evaluates hearing impairment in real-life situations with and without hearing aids. Participants have to rate how often a given statement is true in their daily life, based on the following seven response alternatives: always (99%), almost always (87%), generally (75%), half-the-time (50%), occasionally (25%), seldom (12%) and never (1%). Ease of communication, reverberation, background noise and aversiveness of sounds make up the four subscales of APHAB. In the first three subscales, higher scores suggest less hearing disability, while lower scores indicate less hearing disability in the aversiveness subscale. The APHAB typically requires 10 minutes or less to complete.
Change in the Audio Processor Satisfaction Questionnaire (APSQ) | One month preoperatively and six months post the activation of the speech processor
  The APSQ is a general questionnaire which is designed to assess the handling hearing devices, taking 5 minutes to complete. It assesses the wearing comfort, sound quality, and other device-specific factors related to the audio processor with 15 items on a VAS scale from 0 ('does not agree at all') to 10 ('fully agrees'). If an item does not apply to the subject, then the subject can tick the 'not applicable' option. The maximum number of incomplete answers for the validation analyses is set at three items per subject; if this number exceeds, then the subject shall be excluded. Hence, if participants do not wear at least one hearing device preoperatively, they will only complete in the questionnaire 6 months postactivation.
Change in the Speech, Spatial, and Qualities of Hearing Questionnaire with 12 items (SSQ12) | One month preoperatively and six months post the activation of the speech processor
  The SSQ12 is designed to measure self-reported auditory disability across a wide variety of domains, reflecting the reality of hearing in the everyday world. It takes approximately 5 minutes to complete and it covers: hearing speech in a variety of competing contexts, the directional, distance, and movement components of spatial hearing, segregation of sounds and attending to simultaneous speech streams, ease of listening, the naturalness, clarity, and identifiability of different speakers, different musical pieces and instruments, and different everyday sounds.
  The SSQ12 consists of 12 questions that the subjects score on a scale from 0 (not at all) to 10 (perfectly). The total score is the sum of all items and can range between 0 and 120.
Change in the Hearing Implant Sound Quality Index 19 (HISQUI19) | One month preoperatively and six months post the activation of the speech processor
  The HISQUI19 is a self-administered questionnaire to quantify the individual perceived sound quality of hearing implanted patients in daily life. The questionnaire consists of 19 seven-level Likert items ranging from "always (99%)" to "never (1%)", taking approximately 10 minutes to complete. Added percentage values support the answering. The total score is the sum of all items and ranges from 19 to 133 points. Missing data and the answer option ´not applicable' (N/A) are treated as ´missing values'. The maximum number of incomplete answers are set at three items per subject; if this number exceeds the subject shall be excluded.
Change in Pure tone audiometry | One month preoperatively and six months post the activation of the speech processor
  Pure tone audiometry will be performed according to current clinical standards (ISO 8253-1, 2010) by an experienced Good Clinical Practice (GCP) certificated audiologist (Master of science). Pre- and postoperatively, best-aided pure tone audiometry will be measured at 500, 1000, 2000, 4000 and 8000 Hz using warble tones in sound field in a sound treated booth. The loudspeaker will be placed in front of the participant at ear level at 1 meter distance. The best-aided pure tone average (PTA4) will be calculated by averaging participants' hearing thresholds at 500, 1000, 2000 and 4000 Hz in best-aided condition.
Change in Speech intelligibility | One month preoperatively and six months post the activation of the speech processor
  Speech intelligibility will be evaluated in quiet, using disyllables in Spanish and monosyllables in the other languages, and in noise, using sentences. These tests will be performed pre- and postoperatively in best-aided situation according to current clinical standards (ISO 8253-1, 2010). Participants will be sitting in front of the loudspeaker, positioned at ear level, at a one-meter distance. They will be instructed to repeat the speech stimuli they hear. Speech materials and assessment methods are aligned across the different centers cooperating in this study to obtain comparable results.
Change in Sound localization | One month preoperatively and six months post the activation of the speech processor
  Each center will use its own particular localization set-up. Centers not disposing of an appropriate set-up will only use the SSQ12 spatial subscale. The other centers use both the subjective SSQ12 and the objective localization test.

SECONDARY OUTCOMES:
Change in the Nijmegen Cochlear Implant Questionnaire (NCIQ) | One month preoperatively and six months post the activation of the speech processor
  The NCIQ is a disease-specific measure for QOL and focuses on the needs of CI recipients. It consists of 60 items, taking approximately 15 minutes to complete and it is categorized in the following subdomains: Sound perception basic, Sound perception advanced, Speech production, Self-esteem, Activity and Social interactions. Each subdomain contains 10 items. 55 of the total of 60 items are formulated as statements with 5 answer categories to indicate the degree to which the statement is true: never (1), sometimes (2), often (3), mostly (4), and always (5). The other 5 items will be answered according to the CI user's ability to perform the action in question: no (1), poorly (2), moderate (3), adequate (4), and good (5). If a statement does not apply to a patient, a sixth answer can be given: "not applicable." Missing values and the response category "not applicable" will be both treated as not completed.
Subject demographics | One month preoperatively and six months post the activation of the speech processor
  Subject demographics will be retrieved from the participants' medical file or by asking them if the information is not available. The 11th revision of the International Statistical Classification of Diseases and Related Health Problems (ICD-11) classification will be used to code subjects' health conditions.

CONTACTS AND LOCATIONS:
Locations (5):
- Fiona Stanley Fremantle Hospital Group, Perth, Australia
- University Hospital Antwerp, Edegem, Belgium
- University Clinic of Würzburg, Würzburg, Germany
- World Hearing Centre, Kajetany, Poland
- Hospital La Paz, Madrid, Spain

REFERENCES:
- [Derived] Andries E, Lorens A, Skarzynski PH, Skarzynski H, Calvino M, Gavilan J, Lassaletta L, Tavora-Vieira D, Acharya A, Kurz A, Hagen R, Anderson I, Koinig K, Abdelsamad Y, Van de Heyning P, Van Rompaey V, Mertens G. Impact of cochlear implant indications on outcome, assessed and reported using the international classification of functioning, disability and health model. Eur Arch Otorhinolaryngol. 2025 Oct;282(10):5153-5167. doi: 10.1007/s00405-025-09454-1. Epub 2025 Jun 3. PMID 40456899